CLINICAL TRIAL: NCT03413137
Title: A Prospective Cohort Study Comparing Transperineal to Transrectal MRI-US Fusion Prostate Biopsy
Brief Title: Comparing Transperineal to Transrectal MRI-US Fusion Prostate Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0618-17-RMC
Record Dates: First submitted 2017-10-15; First posted 2018-01-29 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-10

CONDITIONS: Prostate Biopsy
Keywords: Prostate cancer; transperineal mp-MRI-fusion/TRUS biopsies; mp-MRI fusion/TRUS transrectal biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Using the NaviGo™ system each patient will undergo a biopsy using the transperineal followed by transrectal approach.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): A Transperineal mpMRI-US Fusion prostate biopsy followed by a Transrectal mpMRI-US Fusion prostate biopsy
  Interventions: Procedure: Transperineal mpMRI-US Fusion prostate biopsy; Procedure: Transrectal mpMRI-US Fusion prostate biopsy
- Arm B (Active Comparator): A Transrectal mpMRI-US Fusion prostate biopsy followed by a Transperineal mpMRI-US Fusion prostate biopsy
  Interventions: Procedure: Transperineal mpMRI-US Fusion prostate biopsy; Procedure: Transrectal mpMRI-US Fusion prostate biopsy

INTERVENTIONS:
Procedure: Transperineal mpMRI-US Fusion prostate biopsy — mpMRI-US Fusion prostate biopsy in a transperineal approach to direct the needles towards an area in the prostate that was found as suspicious of malignancy by previous MRI imaging, defined as region of interest (ROI).
  Other Names: MRI-US Fusion TP
Procedure: Transrectal mpMRI-US Fusion prostate biopsy — using the same system and MRI imaging, a transrectal approach would be used to sample a few more cores from the ROI as defined by the MRI imaging.
  Other Names: MRI-US Fusion TR

SUMMARY:
This will be a prospective cohort trial that compares transperineal to transrectal MRI-US fusion prostate biopsy

DETAILED DESCRIPTION:
This will be a prospective cohort trial that compares transperineal to transrectal MRI-US fusion prostate biopsy among men. The target population are males that are schedule to undergo MRI-US Fusion prostate biopsy and have an MRI of the prostate. All the pathological samples would be conducted from the area in the prostate that was found as suspicious of malignancy by previous MRI imaging, and defined as region of interest (ROI).

First the prostate biopsy will be preformed in a transperineal approach; Then a transrectal approach would be used to sample a few more cores.

The primary endpoint will be To compare the detection rate for clinically significant prostate cancer between transperineal vs transrectal mp-MRI-fusion/TRUS biopsies. Additionally, the study aims to determine the accuracy of prostate cancer detection in transperineal vs transrectal mp-MRI-fusion/TRUS biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Men who are scheduled to undergo, transrectal or transperineal biopsy and have an MRI of the prostate.

   • Either primary biopsy or repeated biopsy
2. Age 18-90.
3. PI-RADS classification of 3-5

Exclusion Criteria:

1. Men who do not have an MRI of the prostate.
2. PI-RADS classification of 2 or lower
3. Men who were diagnosed with prostate cancer and have begun treatment

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Detection rate for clinically significant prostate cancer | within 2 years
  To compare the detection rate for clinically significant prostate cancer between transperineal vs transrectal mp-MRI-fusion/TRUS biopsies.

SECONDARY OUTCOMES:
Percentage of cores positive per region of interest (ROI) | within 2 years
  To determine the accuracy of prostate cancer detection in transperineal vs transrectal mp-MRI-fusion/TRUS biopsies - Percentage of cores positive per region of interest (ROI)
Amount of volume of cores positive per region of interest (ROI) | within 2 years
  To determine the accuracy of prostate cancer detection in transperineal vs transrectal mp-MRI-fusion/TRUS biopsies - Amount of volume of cores positive per region of interest (ROI)

CONTACTS AND LOCATIONS:
Overall Officials: David Margel, MD PhD, Principal Investigator — Rabn Medical Center, Beilinson Campus
Locations (1):
- Rabin Medical Center, Beilinson campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided